CLINICAL TRIAL: NCT02967302
Title: NEUROIMPA "Intraarticular Application of Opioids in Chronic Arthritis"
Brief Title: NEUROIMPA - Intraarticular Application of Opioids in Chronic Arthritis of the Knee Joint
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hildrun Haibel (Other)
Collaborators: DLR German Aerospace Center (Other)
Responsible Party: Sponsor-Investigator, Hildrun Haibel, Priv. Doz. Dr. med. Hildrun Haibel, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEUROIMPA2015
Record Dates: First submitted 2016-11-10; First posted 2016-11-18 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Knee Arthritis
Keywords: knee arthritis, morphine, local injection, pain
MeSH Terms: conditions — Pain | interventions — Morphine; Triamcinolone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Morphine Sulfate (Experimental): Morphine 3 mg intraarticular once at baseline
  Interventions: Drug: Morphine Sulfate
- Triamcinolone (Active Comparator): Triamcinolone 40 mg intraarticular once at baseline
  Interventions: Drug: Triamcinolone
- Placebo (Placebo Comparator): NaCl 0,9% 5 ml intraarticular at baseline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Morphine Sulfate — active intervention
  Other Names: Morphin Hexal
  Arms: Morphine Sulfate
Drug: Triamcinolone — active control
  Other Names: Triamcinolon Liechtenstein
  Arms: Triamcinolone
Drug: placebo — placebo control
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
To investigate pain and inflammatory parameters (cytokines, immune cells) in knee joint tissue of chronic arthritis patients following intraarticular (i.a.) injections of morphine, a standard steroid or placebo.

The primary hypothesis is that i.a. morphine results in significantly lower pain scores and supplemental analgesic consumption than placebo during the first week after injection, an efficacy comparable to standard i.a. steroid (triamcinolone) medication.

DETAILED DESCRIPTION:
3 arm, double blind, placebo controlled, prospective, mo-nocenter study, which will be conducted in the Department of Rheumatology, Charité University Medicine Berlin, Cam-pus Benjamin Franklin in collaboration with several rheu-matology and orthopedic practices in the Berlin area. Ultra-sound guided synovial needle biopsy and interventions will only be performed at CBF.

Eligible patients will be treated with either morphine 3 mg i.a., NaCl 0.9% i.a. or triamcinolone 40 mg i.a. at Baseline. The entire study period will be 2 weeks per patient.

Assessment of the primary outcome parameter will be at week 1. The patients will be monitored closely throughout the entire study period with a total of 4 visits (screening, baseline, week 1, week 2).

Safety data will be collected in the adverse events form, vital parameters, physical examination and laboratory tests dur-ing the whole study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically detectable and/or ultrasound-visible knee ef-fusion as part of spondyloarthritis (Assessments in SpondyloArthritis international Society, ASAS criteria), Rheumatoid Arthritis, RA (according to American Col-lege of Rheumatology, ACR criteria), undifferentiated mono- or oligoarthritis, Osteoarthritis of the knee, OA.
2. baseline pain score (on a 100 mm Visual Analogue Scale, VAS) >40 mm;
3. male and female patients, age ≥18 - 80 years,
4. body weight 50 - 90 kg.
5. Able and willing to give a written informed consent and comply with the requirements of the study protocol. Only patients who give written informed consent will be in-cluded in the trial.
6. If female: either not of child-bearing potential (meno-pausal since 1 year or surgically sterile) or is willing and able to practice a reliable method of contraception throughout the study with a pearl index <1. Reliable methods of contraception are: condoms plus other methods: implants, injecatbles, combined oral contracep-tives, intrauterine devices, initiated at least 90 days prior to screening. Further reliable methods are a vasecto-mised partner (at least 1 year prior to enrolment), sexual-ly abstinent, surgically sterilized (including hysterecto-my), postmenopausal defined as at least 1 year of spon-taneous amenorrhea (in questionable cases a blood sample with simultaneous levels of follicle stimulating hormone (FSH) above 40 U/l and estradiol below 30 nl/l is confirmatory).
7. If male: either not of child-bearing potential (surgically sterilized, e.g. vasectomy) or is willing and able to prac-tice a reliable method of contraception with a pearl index <1 (see inclusion criterium 6) throughout the study.

Exclusion Criteria:

1. Severe cardiovascular, respiratory, metabolic, neurologi-cal, psychiatric disorders; current bacterial infection es-pecially of the knee
2. abuse of analgesics, benzodiazepines, alcohol; "hard drugs"
3. pregnancy, lactation
4. before biopsy thrombocyte count < 100/nl, Quick <50%
5. intake of anticoagulants, anti-aggregants as monothera-py such as ASS 100 will be allowed
6. participation in an investigational trial during the last 30 days or 5 HLT whichever is longer
7. treatment with intraarticular steroids during the past 4 weeks in the selected joint.
8. Patients with a history of a severe psychiatric illness, which might interfere with the patient's ability to under-stand the requirements of the study and assessment.
9. Patients who are institutionalised due to regulatory or juridical order. Patients who are an employee of the in-vestigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator.
10. Known hypersensitivity to any component of the study medication to morphine or triamcinolone, ileus, respira-tory depression, severe chronic obstructive airway dis-eases, acute abdomen, coagulopathy and/ or infections of the injection site, instability of the injected joint, psori-atic skin manifestation at the injection site, periarticular calcification, non-vascularized bone necrosis, tendon rupture, Charcot-joint.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of pain intensity (on a 100mm VAS) at 8 a.m. on day 7 compared to baseline | 1 week
  Reduction of pain intensity (on a 100mm VAS) at 8 a.m. on day 7 compared to baseline

SECONDARY OUTCOMES:
Area under the VAS curve (AUC) of VAS pain during the first week until 8 p.m. on day 7 | 1 week
  Area under the VAS curve (AUC) of VAS pain during the first week until 8 p.m. on day 7
Pain intensity on McGill pain questionnaire (MPQ) at baseline, week 1 and 2 | 2 weeks
  Pain intensity on McGill pain questionnaire (MPQ) at baseline, week 1 and 2
daily activities at baseline, week 1 and 2 | 2 weeks
  daily activities at baseline, week 1 and 2
activity and mobility of the knee joint (Lysholm Gilquist-Score) at baseline, week 1 and 2 | 2 weeks
  activity and mobility of the knee joint (Lysholm Gilquist-Score) at baseline, week 1 and 2
WOMAC scale (before i.a. injections at baseline, week 1 and 2) | 2 weeks
  WOMAC scale (before i.a. injections and at the end of each week)
nflammatory parameters (cellular infiltrate, opioid receptors and peptides, IL-17, TNFα) in synovial biopsies and fluid (before i.a. medication at baseline and week 1), | 1 weeks
  nflammatory parameters (cellular infiltrate, opioid receptors and peptides, IL-17, TNFα) in synovial biopsies and fluid (before and 7 days af-ter i.a. medication),
supplementary analgesic consumption continuously in the patients diary, recorded at week 1 and 2 | 2 weeks
  supplementary analgesic consumption continuously in the patients diary, recorded at week 1 and 2
Any systemic (e.g. nausea, sedation) and local side effects (infection, tissue injury) will be recorded continuously in the patients diary, recorded at week 1 and week 2. | Screening, Baseline, week 1, week 2
  Any systemic (e.g. nausea, sedation) and local side effects (infection, tissue injury) will be recorded continuously in the patients diary, recorded at week 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Hildrun Haibel, PD Dr, Principal Investigator — Charité CBF, Rheumatology, Berlin, Germany
Locations (1):
- Charité CBF Rheumatology, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
no plan